CLINICAL TRIAL: NCT01019850
Title: Vorinostat With 131-I MIBG Therapy for Resistant/Relapsed Neuroblastoma: A Phase I Study IND# 105,744
Brief Title: N2007-03: Vorinostat and 131-I MIBG in Treating Patients With Resistant or Relapsed Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000659059; P01CA081403 (NIH); N2007-03 (Other: NANT Consortium)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Vorinostat; 3-Iodobenzylguanidine; Peripheral Blood Stem Cell Transplantation; Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment for All Patients (Other): Patients on study will receive vorinostat orally once daily on days 1 to 14. The starting dose level is 180 mg/M2. The maximum dose is 400 mg. Patients will receive 131- I Metaiodobenzylguanidine on day 3, 1hr after vorinostat dosing. Patients will initially receive 8 mCi/kg 131-I MIBG with 180 mg/m2/dose vorinostat. The dose of 131-I MIBG will be escalated in subsequent cohorts to 15 mCi/kg and then to 18 mCi/kg. Peripheral Blood Stem Cell Infusion is planned for 2 weeks after MIBG infusion (day 17). The dose for Purged PBSC is a minimum of 2 x 106 viable CD34+ cells/kg and for Unpurged PBSC: a minimum of 2 x 106 viable CD34+ cells/kg. Stem cells must be infused over 15-30 minutes and within 1.5 hours of thawing. Patients will receive filgrastim following hematopoietic stem cell infusion according to institutional guidelines.
  Interventions: Drug: Vorinostat; Radiation: 131- I Metaiodobenzylguanidine; Procedure: Peripheral Blood Stem Cell Infusion; Drug: Filgrastim

INTERVENTIONS:
Drug: Vorinostat — Patients on study will receive vorinostat orally once daily on days 1 to 14 of treatment.This is a single course treatment. The study has a planned dose escalation schedule, the starting dose level is 180 mg/M2.The maximum absolute dose of vorinostat is 400 mg.
  Other Names: SAHA; Suberoylanili de hydroxamic acid.; Zolinza
Radiation: 131- I Metaiodobenzylguanidine — Patients will receive 131-I MIBG on day 3 , one hour after vorinostat dosing.Patients will initially receive 8 mCi/kg 131-I MIBG with 180 mg/m2/dose vorinostat. The dose of 131-I MIBG will be escalated in subsequent cohorts to 15 mCi/kg and then to 18 mCi/kg.If the starting dose exceeds the maximum tolerated dose, patients will be treated with a lowering of vorinostat dose initially (150 mg/m2/day . Dose level -1). If this combination still exceeds the maximum tolerated dose, then a dose level using reduced dose 131-I MIBG will be studied (6 mCi/kg. Dose level -2).
  Other Names: 131-I MIBG; Iobenguane I 131
Procedure: Peripheral Blood Stem Cell Infusion — Stem cell infusion is planned for 2 weeks after MIBG infusion (day 17). However, stem cells may be infused on day 18 or day 19 to avoid weekend or holiday stem cell infusions.The dose for Purged PBSC is a minimum of 2 x 106 viable CD34+ cells/kg and for Unpurged PBSC: a minimum of 2 x 106 viable CD34+ cells/kg must be available. Stem cells must be infused over 15-30 minutes and within 1.5 hours of thawing.Stem cells will be infused following institutional guidelines for prophylaxis of hypersensitivity reactions and monitoring.
  Other Names: PBSC; Peripheral blood stem cell transplant (PBSCT); Autologous bone marrow transplant (ABMT); Hemopoietic stem cell transplant (HSCT)
Drug: Filgrastim — All patients will receive filgrastim following hematopoietic stem cell infusion according to institutional guidelines (section 4.2.3 of protocol).
  Other Names: G-CSF; Neupogen

SUMMARY:
RATIONALE: Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radioactive drugs, such as iobenguane I 131, may carry radiation directly to tumor cells and not harm normal cells. Giving vorinostat together with iobenguane I 131 may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of giving vorinostat together with iobenguane I 131 in treating patients with resistant or relapsed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of vorinostat in combination with iobenguane I 131 in patients with resistant or relapsed neuroblastoma.
* To define the toxicities of vorinostat in combination with therapeutic doses of iobenguane I 131 in these patients.

Secondary

* To describe, within the context of a phase I study, the response rate in patients treated with vorinostat and iobenguane I 131.
* To describe histone acetylation levels and norepinephrine transporter mRNA levels in peripheral blood mononuclear cells after treatment with different doses of vorinostat.

OUTLINE: This is a multicenter study.

Patients receive oral vorinostat once daily on days 1-14 and iobenguane I 131 IV over 1½-2 hours on day 3. Patients undergo autologous peripheral blood stem cell transplantation on day 17.

Blood samples may be collected periodically for correlative biological studies.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 24 months and no older than 30 years of age when registered on study.
* Patients must have relapsed neuroblastoma, refractory neuroblastoma that had less than a partial response to standard treatment or persistent neuroblastoma that had at least a partial response to standard treatment.
* Patients who have at least a partial response to standard treatment who still have neuroblastoma that can be seen on CT/MRI or MIBG scans must have a surgical biopsy done of the tumor to confirm that it is neuroblastoma. Patients with relapsed or refractory neuroblastoma do not need to have a biopsy done to enter on study.
* Patients must have evidence of MIBG uptake into tumor at one site within 4 weeks prior to entry on study and subsequent to any intervening therapy.
* Patients must have a stem cell product available that meets study criteria. If they don't already have stem cells frozen away then they must be able to have a stem cell collection done to collect the necessary amount of stem cells for study entry and these stem cells must meet study criteria.
* Patients must have adequate heart, kidney, liver and bone marrow function. Patients who have bone marrow disease must meet the bone marrow function criteria to enter the study.

Exclusion Criteria:

* They have had treatment with 131I-MIBG before.
* They have had prior treatment with vorinostat or other HDAC inhibitor.
* They have had a stem cell transplant using another person as the stem cell donor. (You can still be in the study if a previous transplant used your own stem cells)
* They have other medical problems that could get much worse if they had this treatment.
* They are on dialysis for bad kidney function.
* They have a history of unexplained blood clot, pulmonary embolus, thrombotic stroke, or arterial clot.
* They are pregnant or breast feeding.
* They have active infections such as hepatitis or fungal infections.
* They had total body radiation or radiation to the entire belly or a large amount of radiation to the liver or kidney (some radiation to the liver or kidneys is ok).
* They can't cooperate with the special precautions that are needed during MIBG treatment.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
All toxicities , including dose limiting toxicities, of the combination of vorinostat with therapeutic doses of 131-I MIBG | From day 1 of vorinostat therapy to 56 days after stem cell re-infusion
  All toxicities observed will be summarized in terms of type (organ affected or laboratory determination), severity (by NCI CTCAE) and attribution. Tables will be created to summarize these toxicities and side effects by dose level and by course.

SECONDARY OUTCOMES:
Response evaluation , within the context of a phase I study. | At study entry, 56 days after stem cell re-infusion (end of therapy).
  Eligible patients with measurable or evaluable disease who receive 131-I MIBG are evaluable for response even if they fail to complete the course of therapy because of disease progression. Responses will be described for all patients registered on the study even if there are major protocol deviations .
Histone acetylation levels and norepinephrine transported mRNA levels in peripheral blood mononuclear cells after treatment with different doses of vorinostat. | Baseline, Pre-day 3 , Post-day 3, Day 12, 13 or 14.
  Collection of samples for correlative biology is optional and not required for study entry. Although these studies are not mandated, all institutions are strongly urged to submit specimens for all consenting patients.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DuBois, MD, Principal Investigator — UCSF Medical Center at Parnassus
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Salter Packer Children's Hospital, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington